CLINICAL TRIAL: NCT02104765
Title: A Single and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LY2951742 Administered Subcutaneously to Japanese and Caucasian Healthy Subjects
Brief Title: A Study of LY2951742 in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15435; I5Q-MC-CGAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 5 mg LY2951742 Single Dose (Experimental): 5 mg LY2951742 given subcutaneously once
  Interventions: Drug: LY2951742
- 50 mg LY2951742 Single Dose (Experimental): 50 mg LY2951742 given subcutaneously once
  Interventions: Drug: LY2951742
- 120 mg LY2951742 Single Dose (Experimental): 120 mg LY2951742 given subcutaneously once
  Interventions: Drug: LY2951742
- 300 mg LY2951742 Single Dose (Experimental): 300 mg LY2951742 given subcutaneously once
  Interventions: Drug: LY2951742
- 300 mg LY2951742 Multiple Dose (Experimental): 300 mg LY2951742 given subcutaneously once every 4 weeks (Q4W)
  Interventions: Drug: LY2951742
- Placebo Single Dose (Placebo Comparator): Placebo given subcutaneously once
  Interventions: Drug: Placebo
- Placebo Multiple Dose (Placebo Comparator): Placebo given subcutaneously once every 4 weeks (Q4W)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2951742 — Administered subcutaneously.
  Arms: 120 mg LY2951742 Single Dose; 300 mg LY2951742 Multiple Dose; 300 mg LY2951742 Single Dose; 5 mg LY2951742 Single Dose; 50 mg LY2951742 Single Dose
Drug: Placebo — Administered subcutaneously.
  Arms: Placebo Multiple Dose; Placebo Single Dose

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as LY2951742 in healthy Japanese and Caucasians. The study will also investigate how the body processes the drug and how the drug affects the body. The study is expected to last about 5 to 7 months, depending on the arm.

ELIGIBILITY:
Inclusion Criteria:

* Participants are either Caucasian or first generation Japanese.
* Participants' body mass index (BMI) is between 18.0 and 35.0 kilogram per meter square (kg/ m^2).

Exclusion Criteria:

* Participants are heavy caffeine drinkers defined by regular intake of more than 5 cups of coffee (or equivalent in xanthine containing beverages) per day, and/or are unable or unwilling to abide by caffeine restrictions as specified in the protocol.
* Participants are smoking within the previous 6 months.
* Participants have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) prior to dosing or have received a vaccination within 1 month.
* Participants have known allergies to LY2951742, related compounds or any components of the formulation, or history of significant atopy.
* Participants are allergies to either humanized monoclonal antibodies, diphenhydramine, epinephrine, or methylprednisolone.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cypress, California, United States

REFERENCES:
- [Derived] Kielbasa W, Quinlan T. Population Pharmacokinetics of Galcanezumab, an Anti-CGRP Antibody, Following Subcutaneous Dosing to Healthy Individuals and Patients With Migraine. J Clin Pharmacol. 2020 Feb;60(2):229-239. doi: 10.1002/jcph.1511. Epub 2019 Sep 4. PMID 31482569

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (SD): 1 subcutaneous (SC) dose of placebo
- 5 mg LY2951742 Single Dose (SD): 1 SC dose of 5 mg LY2951742
- 50 mg LY2951742 (SD): 1 SC dose of 50 mg LY2951742
- 120 mg LY2951742 (SD): 1 SC dose of 120 mg LY2951742
- 300 mg LY2951742 (SD): 1 SC dose of 300 mg LY2951742.
- Placebo Q4W: 3 SC doses of placebo every 4 Weeks (Q4W)
- 300 mg LY2951742 Q4W: 3 SC doses of 300 mg LY2951742 Q4W
Period: Overall Study
Arm/Group | Placebo (SD) | 5 mg LY2951742 Single Dose (SD) | 50 mg LY2951742 (SD) | 120 mg LY2951742 (SD) | 300 mg LY2951742 (SD) | Placebo Q4W | 300 mg LY2951742 Q4W
Started | 8 | 6 | 6 | 7 | 8 | 2 | 8
Received at Least 1 Dose of Study Drug | 8 | 6 | 6 | 7 | 8 | 2 | 8
Completed | 8 | 6 | 5 | 6 | 7 | 2 | 7
Not Completed | 0 | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (SD) | 5 mg LY2951742 Single Dose (SD) | 50 mg LY2951742 (SD) | 120 mg LY2951742 (SD) | 300 mg LY2951742 (SD) | Placebo Q4W | 300 mg LY2951742 Q4W | Total
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 8 | 2 | 8 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (11.6) | 38.8 (9.9) | 42.7 (12.2) | 34.6 (11.0) | 35.5 (10.3) | NA (NA) — N=2, individual data is 29 and 45 years | 44.8 (11.0) | 40.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 1 | 2 | 3 | 1 | 4 | 19
  Male | 3 | 3 | 5 | 5 | 5 | 1 | 4 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 8 | 6 | 6 | 6 | 8 | 1 | 7 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 3 | 4 | 5 | 1 | 5 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 3 | 3 | 3 | 1 | 3 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 6 | 6 | 7 | 8 | 2 | 8 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section
Time Frame: Baseline through Day 197
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Q4W: 3 SC doses of placebo Q4W
Arm/Group | Placebo (SD) | 5 mg LY2951742 Single Dose (SD) | 50 mg LY2951742 (SD) | 120 mg LY2951742 (SD) | 300 mg LY2951742 (SD) | Placebo Q4W | 300 mg LY2951742 Q4W
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 8 | 2 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2951742
Description: Cmax was evaluated to delineate dose proportionality for the dose cohorts using a power model for geometric means and coefficient of variation. Statistical analysis was not prespecified.
Time Frame: Day 1: Predose, 8 hr and 24 hour postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millliliter (ng/mL)
Groups:
- 5 mg LY2951742 (SD): 1 SC dose of 5 mg LY2951742
Arm/Group | 5 mg LY2951742 (SD) | 50 mg LY2951742 (SD) | 120 mg LY2951742 (SD) | 300 mg LY2951742 (SD) | 300 mg LY2951742 Q4W
Number analyzed (Participants) | 6 | 5 | 7 | 8 | 7
nanogram/millliliter (ng/mL) | 775 (27) | 4270 (58) | 18000 (21) | 41400 (18) | 36300 (42)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve, Zero to Infinity ( AUC[0-∞])
Description: AUC was evaluated to delineate dose proportionality for the dose cohorts using a power model for geometric means and coefficient of variation. Statistical analysis was not prespecified.
Time Frame: Day 1: Predose, 8 hr and 24 hour postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 300 mg LY2951742 Q4W, Day 57: 3 SC doses of 300 mg LY2951742 Q4W
Arm/Group | 5 mg LY2951742 (SD) | 50 mg LY2951742 (SD) | 120 mg LY2951742 (SD) | 300 mg LY2951742 (SD) | 300 mg LY2951742 Q4W, Day 57
Number analyzed (Participants) | 6 | 5 | 7 | 8 | 7
ng*hr/mL | 27600 (24) | 173000 (51) | 733000 (38) | 1520000 (33) | 757000 (41)

ADVERSE EVENTS:
Description: All participants who received at least 1 dose of study drug.
Groups:
- 5 mg LY2951742 Single Dose (SD): 1 SC dose 5 mg of LY2951742
- 50 mg LY2951742 (SD): 1 SC dose 50 mg LY2951742
- 120 mg LY2951742 (SD): 1 SC dose 120 mg of LY2951742
- 300 mg LY2951742 (SD): 2 SC doses 300 mg of LY2951742
Arm/Group | Placebo (SD) | 5 mg LY2951742 Single Dose (SD) | 50 mg LY2951742 (SD) | 120 mg LY2951742 (SD) | 300 mg LY2951742 (SD) | Placebo Q4W | 300 mg LY2951742 Q4W
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/7 | 0/8 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 6/8 | 5/6 | 5/6 | 6/7 | 8/8 | 2/2 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (SD) (N=8) | 5 mg LY2951742 Single Dose (SD) (N=6) | 50 mg LY2951742 (SD) (N=6) | 120 mg LY2951742 (SD) (N=7) | 300 mg LY2951742 (SD) (N=8) | Placebo Q4W (N=2) | 300 mg LY2951742 Q4W (N=8)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 3 (4) | 5 (5) | 4 (4) | 2 (2) | 6 (11) | 2 (5) | 6 (9)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (10)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0/5 (0) | 0/3 (0) | 0/1 (0) | 0/2 (0) | 0/3 (0) | 0/1 (0) | 1/4 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0/5 (0) | 0/3 (0) | 0/1 (0) | 0/2 (0) | 0/3 (0) | 0/1 (0) | 1/4 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days